CLINICAL TRIAL: NCT02570880
Title: Effect of Dough Fermentation Time of Bread on the Glycaemic Index
Acronym: SLOWBREAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beatrice Baumer (Other)
Responsible Party: Sponsor-Investigator, Beatrice Baumer, lecturer, Zurich University of Applied Sciences
Organization: Zurich University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SLOWBREAD-15-1
Record Dates: First submitted 2015-10-02; First posted 2015-10-07 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Glycemic Index (MeSH T483740)
MeSH Terms: interventions — Glycemic Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bread sample vs. glucose solution (Experimental): glycemic index
  Interventions: Other: glycemic index (glucose-solution, bread samples)

INTERVENTIONS:
Other: glycemic index (glucose-solution, bread samples) — All participants will test 2 breads, prepared with different fermentation times of dough, both breads will be tested in duplicate. Methode: International Organization for Standardization / Final Draft International Standard 26642, Food products - Determination of the glycaemic index (GI) and recommendation for food classification

SUMMARY:
This study evaluates the impact of dough fermentation times on the glycaemic index of the ensuing breads.

DETAILED DESCRIPTION:
The worldwide prevalence for non-communicable diseases (NCD) is increasing, nutrition is considered to be one of the main modifiable risk factors. An unhealthy diet leads to obesity, which is a further risk factor for NCDs. Excessive carbohydrates but also the nutritional quality of carbohydrates, can be elements defining "unhealthy diets". The nutritional quality of carbohydrates can be expressed as the glycaemic index.

Fermentation time of bread dough could affect the ensuing bread quality to such an extent that it influences ist glycaemic index. If this hypothesis is confirmed, the process of breadmaking could be optimized in order to offer healthier bread varieties on the market.

ELIGIBILITY:
Inclusion Criteria:

* no known food allergy or intolerance;
* no medications known to affect glucose tolerance (excluding oral contraceptives)
* stable doses of oral contraceptives, acetylsalicylic acid, thyroxin, vitamins and mineral supplements or drugs to treat hypertension or osteoporosis are acceptable.

Exclusion Criteria:

* a known history of diabetes mellitus or the use of antihyperglycaemic drugs or insulin to treat diabetes and related conditions;
* a major medical or surgical event requiring hospitalization within the preceding 3 months;
* the presence of disease or drug(s) which influence digestion and absorption of nutrients;
* the use of steroids, protease inhibitors or antipsychotics
* pregnancy / breastfeeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in postprandial glycemia: Glucose in capillary blood samples over 2 hours (blood samples every 15 minutes), after oral intake of bread samples or glucose-solution (reference) | 2 hours for each sample, 7 samples total, on non consecutive days, over 4 weeks
  a drop of capillary blood will be taken every 15 minutes after ingestion of a bread sample containing 50 g of available carbohydrates

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice E Baumer, MSc, MPH, Principal Investigator — ZHAW, Zurich University of Applied Science, Wädenswil, Switzerland
Locations (1):
- ZHAW, Zurich Univeristy of Applied Sciences, Wädenswil, Canton Zürich, Switzerland